CLINICAL TRIAL: NCT05188482
Title: Complex Treatment Using Vibroacoustic Therapy in a Patient With Co-infection and COVID-19: Case Report.
Brief Title: Using Vibroacoustic Therapy in a Patient With Co-infection and COVID-19
Status: Completed | Type: Observational
Sponsor: Astana Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: MUA
Record Dates: First submitted 2022-01-11; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: SARS CoV 2 Infection
Keywords: periprosthetic joint infection; SARS-CoV-2; co-infections; case report.; vibroacoustic therapy
MeSH Terms: conditions — COVID-19; Coinfection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: vibroacoustic therapy — Vibroacoustic respiratory therapy

SUMMARY:
This article describes a case of successful treatment of a 59-year-old man with sepsis as a result of periprosthetic infection against the background of severe SARS-CoV-2-19, who was hospitalized for 59 days, 57 of which were in the intensive care unit. Vibroacoustic pulmonary therapy, the concept of noninvasive ventilation, syndrome therapy, combination antibiotic therapy taking into account the pathogen and antibiotic sensitivity were used in the treatment.

DETAILED DESCRIPTION:
During the pandemic caused by SARS-CoV-2-19, the whole world faced difficulties. Nevertheless, surgeons had to perform surgical treatment for patients who needed immediate help with a confirmed coronavirus infection [1, 2, 3].

Periprosthetic joint infection is a severe and undesirable consequence after arthroplasty [4, 5]. Patients with coronavirus infection and bacterial infection correlate with an unfavorable outcome [6, 7, 8] The effect of vibroacoustic therapy in the treatment of various conditions has not been sufficiently studied [9, 10]. This clinical case describes the complex therapy of a patient with a periprosthetic infection on the background of SARS-CoV-2 using a vibroacoustic pulmonary device.

ELIGIBILITY:
Inclusion Criteria:

* P/F less 300 torr
* COVID-19 Virus Infection

Exclusion Criteria:

* children
* acute stroke
* acute coronary syndrome
* DVT
* implanted pacemaker
* rib fracture
* infection on chest

Ages: 59 Years to 59 Years | Sex: Male
Age Groups: Adult
Study Population: 59-year-old man with sepsis as a result of periprosthetic infection against the background of severe SARS-CoV-2-19,
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change of time spent on ventilation | 1-2 days
  Changing of the time spent by patients on mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- NATIONAL CENTER Scientific Center of Traumatology and Orthopedics named after Academician Batpenov N.D., Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No